CLINICAL TRIAL: NCT05731089
Title: Pre-Operative Versus Post-Operative Intravitreal Aflibercept Injection for Management of DME in Patients Undergoing Cataract Surgery
Brief Title: IVI Aflibercept Before and After Phaco in DME.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hadi Hospital (Other)
Responsible Party: Principal Investigator, Abeer MohamedSadeck Khattab, consultant of ophthalmology, Al Hadi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVI and phaco
Record Dates: First submitted 2023-02-04; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Macular Edema
Keywords: Aflibercept; cataract; diabetic macular edema
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): Patients in group A were planned to defer the cataract surgery until receiving two injections of Aflibercept at monthly interval, the third injection was then given intra-operatively.
  Interventions: Procedure: Phacoemulsification with IVI of aflibercept
- group B (Active Comparator): Patients in group B were planned to undergo cataract surgery first and received the first injection intra-operatively, then received two post-operative injections with a monthly interval.
  Interventions: Procedure: Phacoemulsification with IVI of aflibercept

INTERVENTIONS:
Procedure: Phacoemulsification with IVI of aflibercept — IVI was either before or after cataract surgery

SUMMARY:
To study whether or not cataract surgery should be deferred until treating the co-existing diabetic macular edema (DME) using intravitreal (IVI) anti-vascular endothelial growth factor (anti-VEGF).

DETAILED DESCRIPTION:
A prospective randomized interventional study included diabetic patients with visually significant cataract and DME. Patients were divided into 2 groups. Group A received three pre-operative intravitreal Aflibercept injections with a monthly interval, the third injection was given intra-operatively. Group B received a single intra-operative injection, and two post-operative injections with a monthly interval. follow up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

- Diabetic patients with visually significant cataract

Exclusion Criteria:

* previous vitreoretinal surgery
* laser or intravitreal injections 6 months prior to the procedure
* intractable glaucom
* active intra-ocular inflammation
* retinal detachment
* vitreous hemorrhage
* epi-retinal membranes
* any other retinal vascular or neuroretinal disease.
* Patients with eventual cataract surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
resolving of macular edema | Sixth month
  change in central macular thickness

SECONDARY OUTCOMES:
Improvement of visual acuity | Sixth month
  measuring of BCVA

CONTACTS AND LOCATIONS:
Locations (1):
- Ahady Hospital, Al Qādisīyah, Hawally, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khattab AM, Hagras SM, Lotfy NM. Pre-operative versus post-operative intravitreal aflibercept injection for management of DME in patients undergoing cataract surgery. Graefes Arch Clin Exp Ophthalmol. 2023 Nov;261(11):3223-3229. doi: 10.1007/s00417-023-06138-6. Epub 2023 Jun 17. PMID 37329361